CLINICAL TRIAL: NCT00471679
Title: Phase I Study of an Ethanol-Lock Strategy to Prevent Central Venous Catheter Infections Among Patients With High-Risk Neuroblastoma
Brief Title: Ethanol-Lock Treatment in Preventing Central Venous Catheter Infections in Patients With High-Risk Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-047; P30CA008748 (NIH); MSKCC-07047
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Ethanol

ARMS (1):
- Ethanol-Lock Treatment (Experimental): Ethanol instillation and removal will be carried out by one of the investigating physicians, a pediatric surgical nurse practitioner, or a dedicated research nurse. Syringes containing a 70% ethanol solution will be pre-filled in the PDH pharmacy and dispensed to the nurse caring for a particular patient. The volume of ethanol to be administered into each lumen of the central line will be specific to each patient's catheter and will be determined at enrollment.
  Interventions: Drug: ethanol

INTERVENTIONS:
Drug: ethanol

SUMMARY:
RATIONALE: Ethanol-lock treatment may help prevent central venous catheter infections in patients with high-risk neuroblastoma.

PURPOSE: This phase I trial is studying the side effects of ethanol-lock treatment in preventing central venous catheter infections in patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of the ethanol-lock strategy (ETL) in preventing central venous catheter infections in patients with high-risk neuroblastoma being treated on clinical trial MSKCC-03077.

Secondary

* Determine whether this strategy increases the likelihood of remaining infection-free for 6 months.
* Determine the cumulative incidence of a single positive centrally-drawn blood culture in these patients and compare to previously obtained historical controls.
* Determine the median time-to-infection of the central line, where infection is defined as any positive centrally-drawn (from the treated line) blood culture.
* Determine the cumulative incidence of central line removals in these patients and compare to historical controls.
* Collate the types of organisms among these patients who develop a positive centrally-drawn blood culture and compare to historical controls.

OUTLINE: This is a prospective, nonrandomized, open-label, historical control study.

Patients receive monoclonal antibody 3F8 on clinical trial MSKCC-03077. In each course of monoclonal antibody 3F8 treatment, patients receive ethanol-lock treatment on days 0-3 (after each monoclonal antibody 3F8 infusion) for up to 6 months for central venous catheter management.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma by histopathology OR bone marrow metastases and high urine catecholamine levels

  * High-risk disease
* Currently enrolled on clinical trial MSKCC-03077

  * Expected duration of therapy ≥ 6 months
* Surgically-implanted central venous catheter with documented patency

  * Must be able to establish patency of central venous catheter lumen
* No history of culture-positive central venous catheter infection in catheter to be treated

PATIENT CHARACTERISTICS:

* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN
* No history of hypersensitivity to ethanol
* No history or documented active seizure disorder
* No documented acute liver failure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent total parenteral nutrition or other infusion requiring use of the central line at night
* No concurrent levetiracetam or other anticonvulsants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 2 years

SECONDARY OUTCOMES:
Efficacy, in terms of 6-month infection-free rate, cumulative incidence of infection, cumulative incidence of central line removal, and median time to infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark L. Kayton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Michael P. LaQuaglia, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States